CLINICAL TRIAL: NCT04116034
Title: Alfapump DSR System in the Treatment of Diuretic Resistant Heart Failure Subjects
Brief Title: Alfapump Direct Sodium Removal (DSR) Feasibility Study
Acronym: RED DESERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sequana Medical N.V. (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019-CHF-005
Record Dates: First submitted 2019-10-01; First posted 2019-10-04 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure; Congestive Heart Failure; Cardiorenal Syndrome; Volume Overload; Sodium Excess; Sodium Disorder
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome; Edema; Hypernatremia

STUDY DESIGN:
Intervention Model Description: up to 10 subjects will be enrolled to evaluate feasibility and safety of thealfapump DSR system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DSR (Experimental): Up to 10 subjects will be treated with alfapump DSR system for a total treatment period of 59 days post-implantation
  Interventions: Device: alfapump DSR system

INTERVENTIONS:
Device: alfapump DSR system — Infusion of sodium free Dextrose 10% into peritoneal cavity to remove sodium and fluid using principles of peritoneal dialysis, sodium and ultrafiltrate will be evacuated to the bladder by the alfapump

SUMMARY:
First in Human feasibility and sfafety study of the alfapump DSR system in the treatment of Heart failure subects resistant to diuretic therapy. Up to 10 subjects will be enrolled in up to 3 centres in Belgium and Georgia and will be iplanted with the alfapump DSR system. Subjects will undergo DSR titration during a 2 week hospitalisation period, and will continue titrated DSR therapy as outpatients for 4 more weeks.

DETAILED DESCRIPTION:
Up to 10 subjects diagnosed with stable chronic heart failure (CHF) on high oral diuretic dose and an MDRD eGFR > 30ml/min/1.73m2 will undergo subcutaneous implantation of the alfapump DSR system (Day-13) and portacath system and participate in a 6 week interventional study. Prior to an inpatient study period, the subject will undergo a 40mg IV furosemide (or 1 mg IV bumetanide) diuretic challenge with timed biospecimen collection. On day 14 post-implant (Day 0), the subject will be admitted for a 14-day period in which diuretics will be withheld and subjects will be on a strict low-sodium (3g/day) diet with strict intake/output and all urine collected and samples saved for analysis. During the first 7 days (Day 0 - 6) subjects will be treated with 1000ml of DSR Infusate Monday, Wednesday, Friday administered to the peritoneal cavity through the subcutaneous peritoneal catheter. The infusate will remain in the peritoneal cavity for a 2 hour dwell time, then all fluid will be removed from the peritoneal cavity to the urinary bladder using the alfapump DSR system over the subsequent 8 hours. On day 7, subjects will be transitioned to a moderate to high salt diet given as the same low-sodium (3g/day) diet with supplementation with sodium chloride tablets (2g/day) (5g/day total sodium), as this will likely represent their typical home sodium intake. During this time, the optimal treatment protocol (frequency of administration and volume of DSR infusate administered) for individual subjects based on daily sodium balance, weight changes, and blood pressure will be created and tested over the next seven days in hospital (Day 7 - 13). Following the inpatient period, a second diuretic challenge will be conducted. Over the subsequent 28 days, diuretics will continue to be withheld with preferential maintenance of euvolemia through DSR and subjects will come into the clinic based on their tailored therapy schedule and undergo supervised DSR infusate administration. Addition of diuretic treatment will only be allowed if maximal DSR therapy has been instituted (DSR 7 days per week (i.e., including weekends) at 1.5L per session with dwell time of 4 hours) and/or holding diuretics until additional DSR can be utilized would represent a risk to the subject, as described in the CIP diuretic algorithm.

After the completion of the study period, the alfapump DSR therapy is halted and the subject undergoes a third diuretic challenge to quantify diuretic response. At this point oral diuretic therapy will be resumed. At the end of the study the alfapump can remain implanted and set to 'dormant' state after discussion and agreement between subject and investigator, and if there are no clinical, ethical or other reasons indicating explanation of the alfapump. Alternatively, the subject may elect to enroll into a low intensity follow-on study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects > 18 years of age
2. eGFR > 30ml/min/14.73m2
3. Diagnosis of heart failure with one of the following: a. nt-proBNP > 400 pg/ml (or BNP > 100 pg/mp) and oral diuretic dose ≥ 80mg furosemide (or 20mg torsemide or 1mg bumetanide) OR b. Oral diuretic dose ≥ 120mg furosemide (or 30 mg torsemide or 1.5 mg bumetanide)
4. Stable diuretic dose for 30 days
5. Systolic blood pressure ≥ 100 mmHg
6. Determined by treating provider to be at optimal volume status

Exclusion Criteria:

Candidates for participation will be ineligible for the study if any of the following exclusion criteria apply:

1. Proteinuria > 1g/day
2. BMI > 40
3. History of abdominal surgery or peritonitis
4. Anemia with hemoglobin < 8g/dL
5. Serum sodium < 135 mEq/L
6. Severe hyperkalemia or baseline plasma potassium > 4.5 mEq/L
7. Significant other organ disease or comorbidities
8. Hospitalization within 90 days
9. Cirrhosis
10. Hemodynamically significant stenotic valvular disease
11. Active or recurrent urinary tract infection or history of renal transplant
12. History of significant bladder dysfunction expected to interfere with ability of subject to tolerate DSR pumping into bladder
13. Uncontrolled diabetes with frequent hyperglycemia or Type 1 diabetes
14. Subject is currently participating in another clinical trial
15. Subject is unable to comply with all required study follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Safety in-hospital - Device related | Through Day 14 of treatment period
  Rate of device related serious adverse events
Safety in-hospital - therapy related | Through Day 14 of treatment period
  Rate of therapy related serious adverse events
Safety in-hospital - procedure related | Through Day 14 of treatment period
  Rate of procedure related serious adverse events
Safety during treatment period - device related | through Day 42 of treatment period
  Rate of device related serious adverse events
Safety during treatment period - procedure related | through Day 42 of treatment period
  Rate of procedure serious adverse events
Safety during treatment period - therapy related | through Day 42 of treatment period
  Rate of therapy related serious adverse events

SECONDARY OUTCOMES:
Feasibiity endpoint sodium balance in-hospital | through Day 14 of DSR therapy
  Number of patients with neutral sodium balance (sodium intake equal to sodium output) in the absence of diuretic therapy during hospitalization period
Feasibility endpoint sodium balance during treatment period | Through Day 42 of DSR Therapy
  Number of patients with neutral sodium balance (sodium intake equal to sodium output) in the absence of diuretic therapy in a titrated schedule during treatment period

OTHER OUTCOMES:
Bioimpedance | At baseline, day 7, 14, and 42
  Change in bioimpedance from baseline through treatment
Hemoconcentration markers | At baseline, day 7, 14, and 42
  Change in hemoglobin versus hematocrit ratio from baseline through treatment
N-Terminal Prohormone of Brain Natriuretic Peptide (nt-ProBNP) | At baseline, day 7, 14, and 42
  Change in nt-proBNP from basline through treatment
Weight | At baseline, day 7, 14, and 42
  Change in Weight from baseline through treatment
Glycolated Hemoglobine (HbA1c) | At baseline, day 7, 14, and 42
  Changes in HBA1c from baseline through treatment
Sodium balance | Up to day 42
  Daily sodium balance
Fluid balance | Up to day 42
  Daily fluid balance
6-hour diuretic response | At baseline, day 14, day 42
  Change in response to 6 hour diuretic challenge from baseline through treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Bartunek, MD, Principal Investigator — Onze Lieve Vrouw Hospital Aalst, Belgium
Locations (2):
- OLV Ziekenhuis, Aalst, Belgium
- Tbilisi Heart & Vascular Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No
No IPD data will be shared with other researchers

REFERENCES:
- [Derived] Rao VS, Ivey-Miranda JB, Cox ZL, Moreno-Villagomez J, Ramos-Mastache D, Neville D, Balkcom N, Asher JL, Bellumkonda L, Bigvava T, Shaburishvili T, Bartunek J, Wilson FP, Finkelstein F, Maulion C, Turner JM, Testani JM. Serial direct sodium removal in patients with heart failure and diuretic resistance. Eur J Heart Fail. 2024 May;26(5):1215-1230. doi: 10.1002/ejhf.3196. Epub 2024 Mar 31. PMID 38556717